CLINICAL TRIAL: NCT04081168
Title: COLLISION XL: Unresectable Colorectal Liver Metastases: Stereotactic Body Radiotherapy vs. Microwave Ablation - a Phase II Prospective Randomized Controlled Trial for Intermediate-size (3 - 5 cm) Colorectal Liver Metastases
Brief Title: COLLISION XL: Unresectable Colorectal Liver Metastases (3-5cm): Stereotactic Body Radiotherapy vs. Microwave Ablation
Acronym: COLLISION-XL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Dr. M.R. Meijerink, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL68326.029.19
Record Dates: First submitted 2019-08-27; First posted 2019-09-09 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer Metastatic; Liver Metastasis Colon Cancer
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Stereotactic Body Radiotherapy vs. Microwave Ablation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stereotactic Body Radiotherapy (Active Comparator): Patients included will undergo Stereotactic Body Radiotherapy (SBRT) of hepatic metastases.
  Interventions: Device: Stereotactic Body Radiotherapy
- Microwave Ablation (Active Comparator): Patients included will undergo Microwave Ablation (MWA) of hepatic metastases.
  Interventions: Device: Microwave Ablation

INTERVENTIONS:
Device: Stereotactic Body Radiotherapy — Patients will undergo Stereotactic Body Radiotherapy (SBRT)
  Other Names: SBRT
  Arms: Stereotactic Body Radiotherapy
Device: Microwave Ablation — Patients will undergo Microwave Ablation (MWA)
  Other Names: MWA
  Arms: Microwave Ablation

SUMMARY:
Multiple articles report that thermal ablation is a safe and effective treatment for unresectable colorectal liver metastases (CRLM) ≤3cm. However efficacy of thermal ablation decreases with increasing lesion size. Guidelines state that thermal ablation is the preferred option for unresectable CRLM ≤3cm and stereotactic body radiotherapy (SBRT) when thermal ablation is not possible. It remains uncertain what local treatment method should be recommended for unresectable CRLM of 3-5cm.

DETAILED DESCRIPTION:
Objective: The primary objective of this study is to compare efficacy of MWA to the efficacy of SBRT with regards to the primary endpoint (local tumour progression free survival at 1 year [1-year LTPFS]) in patients with unresectable CRLM (3 - 5 cm) that are unsuitable for surgery due to either comorbidities, a history of extensive abdominal surgery, a poor performance status or due to a certain unfavourable anatomical location of the tumour.

Study design: COLLISION XL is a prospective multi-centre phase-II randomized controlled trial.

Study population: 68 patients with 1-3 unresectable lesions of 3 - 5cm, unsuitable for (further) chemotherapy regimens, suitable for both MWA and SBRT and no or limited extrahepatic disease (1 extrahepatic lesion is allowed, not including positive para-aortal lymph nodes, celiac lymph nodes, adrenal metastases, pleural carcinomatosis or peritoneal carcinomatosis) are considered eligible. Supplementary resections for resectable lesions and thermal ablations for unresectable CRLM ≤3cm are allowed. A maximum number of 10 CRLM are allowed for patients with no extrahepatic disease and a maximum number of 5 lesions are allowed for patients with limited extrahepatic disease.

Intervention: SBRT or MWA. The panel, consisting of at least two interventional radiologists, two hepatobiliary surgeons and two radiation oncologists, will appoint lesions of 3-5cm that are unresectable and suitable for both MWA and SBRT, as target lesions. All lesions that are not suitable for ablation should be resectable and all unresectable lesions <3cm should be suitable for thermal ablation.

Main study parameters/endpoints: Primary endpoint is local tumour progression free survival (LTPFS) at 1 year from randomization. Secondary endpoints are local tumour progression free survival time, OS, disease-free survival (DFS), time to progression (TTP), procedural morbidity/toxicity and mortality, assessment of pain and quality of life (QoL) and cost-effectiveness ratio (ICER).

ELIGIBILITY:
Inclusion Criteria:

* 1-3 unresectable CRLM size 3-5 cm eligible for both MWA and SBRT (target lesions);
* Additional CRLM are allowed if considered either resectable or ablatable and <3cm
* No or limited extrahepatic disease (1 extrahepatic lesion is allowed, not including positive para-aortal lymph nodes, celiac lymph nodes, adrenal metastases, pleural carcinomatosis or peritoneal carcinomatosis);
* For subjects with liver only disease the maximum number of CRLM is 10; for subjects with limited extrahepatic disease the maximum number of CRLM is 5;
* Prior focal liver treatment is allowed
* Subjects without prior focal liver treatment should be either unsuitable for 1st line chemotherapy or have progressed under/after 1st-line chemotherapy;
* Subjects with recurrent (either local or distant-hepatic) CRLM after previous focal treatment should be unsuitable for (further) systemic therapy (further downsizing or conversion to resectable disease improbable).

Exclusion Criteria:

* Compromised liver function (e.g. signs of portal hypertension, INR > 1,5 without use of anticoagulants, ascites);
* Pregnant or breast-feeding subjects;
* Immunotherapy ≤ 6 weeks prior to the procedure;
* Chemotherapy ≤ 6 weeks prior to the procedure;
* Severe allergy to contrast media not controlled with premedication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
One-year local tumor progression-free survival | 1 year
  One-year local tumor progression-free survival

SECONDARY OUTCOMES:
Timo-to-local tumor progression | 5 years
  Timo-to-local tumor progression
Overall survival (OS) | 5 years
  Overall survival (OS)
Disease-Free Survival (DFS) | 5 years
  Disease-Free Survival (DFS)
Mortality | 5 years
  Mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van der Lei S, Dijkstra M, Nieuwenhuizen S, Schulz HH, Vos DJW, Versteeg KS, Buffart TE, Swijnenburg RJ, de Vries JJJ, Bruynzeel AME, van den Tol MP, Scheffer HJ, Puijk RS, Haasbeek CJA, Meijerink MR; and COLLISION Trial Group. Unresectable Intermediate-Size (3-5 cm) Colorectal Liver Metastases: Stereotactic Ablative Body Radiotherapy Versus Microwave Ablation (COLLISION-XL): Protocol of a Phase II/III Multicentre Randomized Controlled Trial. Cardiovasc Intervent Radiol. 2023 Aug;46(8):1076-1085. doi: 10.1007/s00270-023-03498-8. Epub 2023 Jul 10. PMID 37430016